CLINICAL TRIAL: NCT06479772
Title: Evaluation of the Potential Impact of an Artificial Intelligence Solution in Second Reading of Organized Screening.
Acronym: ELIAS
Status: Completed | Type: Observational
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Collaborators: Vivactis M2Research (Industry)
Responsible Party: Sponsor
Other Study IDs: 2021-06-051
Record Dates: First submitted 2023-12-15; First posted 2024-06-28 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Breast Cancer Female

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Based on data from a series of patients who underwent screening mammography with a "normal" or "benign" first-reading result. The main objective of the study is to evaluate the possibilities of subtracting from the second reading of breast cancer screening a population of examinations for which the risk of discovering cancer is close to zero, using an AI system (here the MammoScreen™ system).

DETAILED DESCRIPTION:
This is a retrospective multicenter study of mammography imaging data contained in the PACS (Picture Archiving and Communication System) of six radiology centers located in the Rhône, Puy de dôme, Cantal and Haute-Loire départements.

In order to be able to collect two-year follow-up data, the files analyzed will concern all women who received a screening mammogram during the years 2015, 2016, 2017, 2018 and 2019. More recent mammograms will be excluded.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 50 to 74 participating in the organized screening campaign.
* Having had a screening mammogram with a final L1 result of "normal" (ACR 1/ BI-RADS 1) or "benign" (ACR 2/ BI-RADS 2).
* For which a second reading interpretation is available
* Screening mammograms performed during the years 2015 to2019 (In order to have follow-up data (subsequent mammogram or information on the person's future)

Exclusion Criteria:

- Mammography not performed as part of organized screening

Ages: 50 Years to 74 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female breast cancer
Study Population: As this was a retrospective exploratory study, with no prior hypothesis, the number of subjects required was not calculated.
  The study population (n=55,000) represents, for the radiology practices concerned, all mammograms examined in second reading by the Auvergne Rhône Alpes regional cancer screening coordination center between 2015 and 2019.
Sampling Method: Non-Probability Sample
Enrollment: 55589 (Actual)
Dates: Start 2023-10-10 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Percentage of real negatives | Week 8
  Percentage of cases negatived by MammoScreen (considered benign by the system), and for which no cancer was detected at the end of the L2 (according to the different risk levels of the MammoScreen software - score from 1 to 10). We distinguish two sub-populations: L2- and L2+ with BDD- (in addition to L2-).

SECONDARY OUTCOMES:
Percentage of real positives | Week 8
  Percentage of MammoScreen-positive cases for which cancer was detected in L2 (according to the different risk levels of the MammoScreen software - score from 1 to 10).
Percentage of false negatives | Week 8
  Percentage of MammoScreen-positive cases with an L2 ultimately considered negative (L2- or L2 + with DBB-), for which interval cancer is detected (according to the different risk levels of the MammoScreen software - score from 1 to 10).

CONTACTS AND LOCATIONS:
Overall Officials: Christophe TOURASSE, MD, Principal Investigator — Hôpital Privé Jean Mermoz
Locations (1):
- Hôpital Privé Jean Mermoz, Lyon, France